CLINICAL TRIAL: NCT01845025
Title: A 26 Week, Randomized, Active-controlled Safety Study of Double-blind Formoterol Fumarate in Free Combination With an Inhaled Corticosteroid Versus an Inhaled Corticosteroid in Adolescent and Adult Patients With Persistent Asthma.
Brief Title: Study of Safety of Foradil in Patients With Persistent Asthma
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to the action to withdraw the Foradil Aerolizer NDA in US; study was discontinued. This was a commercial reason and not due to any change in benefit-risk.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CFOR258D2416; 2012-004854-27 (EudraCT Number)
Record Dates: First submitted 2013-04-22; First posted 2013-05-03 (Estimated); Results first posted 2017-03-21 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-01

CONDITIONS: Persistent Asthma
Keywords: Asthma; formoterol fumarate; Foradil; inhaled corticosteroid; fluticasone propionate; safety
MeSH Terms: conditions — Asthma | interventions — Formoterol Fumarate; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FOM 12 mcg + FP (Experimental): Formoterol 12 mcg + fluticasone propionate 100 mcg, 250 mcg or 500 mcg for inhalation
  Interventions: Drug: Formoterol 12 mcg; Drug: Fluticasone propionate 100 mcg; Drug: Fluticasone propionate 250 mcg; Drug: Fluticasone propionate 500 mcg
- fluticasone propionate (FP) (Active Comparator): fluticasone propionate 100 mcg, 250 mcg or 500 mcg + Placebo to Match Formoterol 12 mcg for inhalation
  Interventions: Drug: Fluticasone propionate 100 mcg; Drug: Fluticasone propionate 250 mcg; Drug: Fluticasone propionate 500 mcg; Drug: Placebo

INTERVENTIONS:
Drug: Formoterol 12 mcg — Formoterol 12 mcg one inhalation twice daily, via dry powder inhaler
  Other Names: FOR258
  Arms: FOM 12 mcg + FP
Drug: Fluticasone propionate 100 mcg — Fluticasone propionate 100 mcg one inhalation twice daily via dry powder inhaler
Drug: Fluticasone propionate 250 mcg — Fluticasone propionate 250 mcg one inhalation twice daily via dry powder inhaler
Drug: Fluticasone propionate 500 mcg — Fluticasone propionate 500 mcg, one inhalation twice daily via dry powder inhaler
Drug: Placebo — Placebo to match formoterol one inhalation twice daily via dry powder inhaler
  Arms: fluticasone propionate (FP)

SUMMARY:
The purpose of this study was to assess whether the risk of serious asthma-related events (asthma-related hospitalizations, asthma related intubations, and asthma related deaths) in adolescents and adults (12 years of age and older) taking inhaled formoterol fumarate/fluticasone propionate combination was the same as those taking inhaled fluticasone propionate alone.

DETAILED DESCRIPTION:
This was a 26 week, double blind, randomized, active-controlled safety study of Foradil in free combination with inhaled corticosteroid versus an inhaled corticosteroid alone in adults and adolescent patients with persistent asthma. The primary objective of the study was to demonstrate that the addition of formoterol fumarate to fluticasone propionate is non-inferior to fluticasone propionate alone in terms of the risk of composite serious asthma related events (asthma-related hospitalization, asthma-related intubation, and asthma-related death). The individual components of the composite primary endpoint (i.e., asthma-related hospitalization, asthma-related intubation and asthma-related death) will be assessed as a secondary safety endpoints.

The efficacy assessment is the secondary objective.

ELIGIBILITY:
Key Inclusion Criteria:

1. Written informed consent, and assent if applicable, must be obtained before any assessment is performed.
2. Male or female patients 12 years of age and older
3. Confirmed diagnosis of persistent asthma, as defined by national and international asthma guidelines (e.g., GINA; NIH; etc.) for at least 1 year prior to study enrollment.
4. PEF≥50% of predicted normal value.
5. Current and appropriate use of one of the treatments listed in the protocol for asthma.
6. Recent asthma exacerbation between 30 days and 12 months prior to randomization that either:

   * required treatment with systemic corticosteroids (tablets, suspension, or injection) or
   * required hospitalization (defined as an inpatient stay or >24-hour stay in an observation area in an emergency room or other equivalent facility)

Key Exclusion Criteria:

1. History of life-threatening asthma episode that required intubation and/or was associated with hypercapnia requiring non-invasive ventilatory support.
2. Current evidence of pneumonia, pneumothorax, atelectasis, pulmonary fibrotic disease, allergic bronchopulmonary aspergillosis, cystic fibrosis, bronchopulmonary dysplasia, or other respiratory abnormalities other than asthma.
3. Current evidence of, or past physician assessment of, chronic bronchitis, emphysema, or chronic obstructive pulmonary disease.
4. History of smoking ≥ 10 pack years.
5. Exercise induced asthma (as the only asthma-related diagnosis) not requiring daily asthma control medicine.
6. Suspected or documented bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear that is not resolved at randomization.
7. Worsening/Unstable asthma within 7 days prior to randomization.
8. Any asthma exacerbation requiring systemic corticosteroids within 30 days of randomization or more than 4 separate exacerbations in the 12 months preceding randomization.
9. Two or more hospitalizations for greater than 24 hours duration for treatment of asthma in the 12 months preceding randomization.
10. History of hypersensitivity to any beta2-agonist, sympathomimetic drug, inhaled corticosteroids, or systemic corticosteroid therapy or any component of the possible study treatments in this trial, including severe milk protein hypersensitivity.
11. Use of anti-IgE (e.g., omalizumab) or any other monoclonal antibody, in the 6 months prior to randomization.
12. Use of (Beta) β-blockers within 1 day prior to first dose of study medication.
13. Use of ICS, LABA, ICS+LABA, LTRAs, leukotriene modifiers, anticholinergics, or theophylline must be discontinued prior to the first dose of investigational treatment.
14. Use of a potent CYP3A4 inhibitor within 4 weeks of randomization (e.g., ritonavir, atazanavir, clarithromycin, indinavir, itraconazole, nefazodone, nelfinavir, saquinavir, ketoconazole, telithromycin).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 827 (Actual)
Dates: Start 2013-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chrsitopher Compton, Study Director — Novartis Pharmaceuticals
Locations (24):
- United States (24):
  - Novartis Investigative Site, Avondale, Arizona
  - Novartis Investigative Site, North Hollywood, California
  - Novartis Investigative Site, Bradenton, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Conyers, Georgia
  - Novartis Investigative Site, Stone Mountain, Georgia
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Covington, Louisiana
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Gaithersburg, Maryland
  - Novartis Investigative Site, Picayune, Mississippi
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, North Massapequa, New York
  - Novartis Investigative Site, Elizabeth City, North Carolina
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Oaks, Pennsylvania
  - Novartis Investigative Site, East Greenwich, Rhode Island
  - Novartis Investigative Site, Mt. Pleasant, South Carolina
  - Novartis Investigative Site, Memphis, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, St. George, Utah
  - Novartis Investigative Site, Mequon, Wisconsin
  - Novartis Investigative Site, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Following the decision to stop further enrollment into the study, 1121 patients had been screened, of whom 825 were randomized. Of the 820 patients randomized and treated and part of Intent To Treat (ITT analysis) 5 patients were randomized but were excluded from the ITT analyses as they did not take study medication.
Pre-assignment Details: 827 actual in the protocol section came from the IRT because 2 patients were randomized twice but only counted once.
Period: Overall Study
Arm/Group | FOM 12 mcg + FP | Fluticasone Propionate (FP)
Started | 411 | 409
Completed | 326 | 332
Not Completed | 85 | 77
Not completed — Adverse Event | 6 | 3
Not completed — Unsatisfactory therapeutic effect | 4 | 2
Not completed — Withdrawal by Subject | 48 | 44
Not completed — Lost to Follow-up | 13 | 13
Not completed — Administrative problems | 8 | 8
Not completed — Death | 2 | 0
Not completed — Protocol deviation | 3 | 6
Not completed — Missing | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FOM 12 mcg + FP | Fluticasone Propionate (FP) | Total
Number analyzed (Participants) | 411 | 409 | 820
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (16.67) | 45.6 (17.02) | 45.2 (16.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 284 | 272 | 556
  Male | 127 | 137 | 264

OUTCOME MEASURES:

1. Primary Outcome: Number of First Occurrence(s) of Any Composite Endpoint Including Asthma-related Hospitalizations, Intubations and Deaths During the Study at 26 Weeks
Description: The primary safety endpoint was the number of first occurrence(s) of any composite endpoint. The composite events include asthma-related deaths, asthma-related intubations and asthma-related hospitalizations. The number of events includes all adjudication confirmed events, one patient could experience multiple events during the course of study; Event rate = 100 * n patients with any events / total N patients in treatment group.
Time Frame: 26 weeks
Population: Intent to treat (ITT) population included all randomized patients who took at least one dose (one inhalation) of study medication
Measure: Number; unit: number of occurences
Arm/Group | FOM 12 mcg + FP | Fluticasone Propionate (FP)
Number analyzed (Participants) | 411 | 409
number of occurences
  Composite event | 3 | 3
  Asthma-related death | 0 | 0
  Asthma-related intubation | 0 | 0
  Asthma-related hospitalization | 3 | 3

2. Secondary Outcome: Number of Asthma Exacerbations at 26 Weeks
Description: Number of asthma exacerbations events
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: events
Arm/Group | FOM 12 mcg + FP | Fluticasone Propionate (FP)
Number analyzed (Participants) | 411 | 409
events | 1.3 (0.62) | 1.2 (0.51)

3. Secondary Outcome: Percentage of Days of School/Work Missed at 26 Weeks
Description: The percentage of days of school/work missed during the treatment period (26 weeks). Overall percentage of school days missed for each student patient or of work days missed is calculated by total number of days missed divided by total days of treatment.
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | FOM 12 mcg + FP | Fluticasone Propionate (FP)
Number analyzed (Participants) | 411 | 409
percentage of days | 0.97 (4.558) | 0.56 (1.641)

4. Secondary Outcome: Percentage of Days With Limited Ability to Perform Normal Daily Activities at 26 Weeks
Description: The percentage of days with limited ability to perform normal daily activities during the treatment period (26 weeks). Percentage is calculated as total number of days when the patient had limited ability to perform normal daily activities divided by total days of treatment.
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | FOM 12 mcg + FP | Fluticasone Propionate (FP)
Number analyzed (Participants) | 411 | 409
percentage of days | 4.73 (12.774) | 4.75 (12.705)

5. Secondary Outcome: Percentage of Days With Nighttime Awakenings at 26 Weeks
Description: Percentage of days with nighttime awakenings during the treatment period (26 weeks)
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | FOM 12 mcg + FP | Fluticasone Propionate (FP)
Number analyzed (Participants) | 411 | 409
percentage of days | 4.55 (9.577) | 4.20 (8.956)

6. Secondary Outcome: Percentage of Days With no Rescue Medication Use at 26 Weeks
Description: Percentage of rescue free days is calculated as total number of days with no rescue medication was taken divided by total days of treatment.
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | FOM 12 mcg + FP | Fluticasone Propionate (FP)
Number analyzed (Participants) | 411 | 409
percentage of days | 76.97 (27.255) | 73.29 (30.640)

7. Secondary Outcome: Percentage of Days With no Symptoms at 26 Weeks
Description: Percentage of days with no symptoms during the treatment period (26 weeks). Percentage is calculated as total number of days with no symptoms divided by total days of treatment.
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | FOM 12 mcg + FP | Fluticasone Propionate (FP)
Number analyzed (Participants) | 411 | 409
percentage of days | 79.47 (25.501) | 77.64 (28.394)

8. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ - 6) Total Score at Week 26
Description: Change from baseline in Asthma control Questionnaire (ACQ - 6) total score at week 26. Results of the Asthma control questionnaire (ACQ-6); The average score of the six questions is calculated as the sum of scores divided by the number of questions that were answered at the time point, as long as there were at least 4 questions answered. The ACQ6 score is calculated as the mean of the responses to the first 6 questions of the ACQ. The ACQ is a scale containing 7 questions, each question has a 7-point scale which ranges from 0 to 6; a total score of 0 corresponds to no impairment and a total score of 6 corresponds to maximum impairment.
Time Frame: baseline and 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: total score on a scale
Arm/Group | FOM 12 mcg + FP | Fluticasone Propionate (FP)
Number analyzed (Participants) | 411 | 409
total score on a scale | -0.65 (1.224) | -0.59 (1.094)

9. Secondary Outcome: Unplanned Healthcare Utilization at Visit 3 (Week 4), Visit 4 (Week 12) and Visit 5 (Week 26)
Description: Unplanned healthcare utilization by visit (Telephone contact with study doctor (MD); Telephone contact with other physician (MD) or healthcare provider (HCP); Unscheduled or unplanned visit to study doctor (including home visits); Unscheduled or unplanned visit to other physician or healthcare provider (including home visits); Emergency department or hospital visit (< 24 hours); Hospital admission or Emergency department visit (> 24 hours).
Time Frame: Week 4, Week 12, and Week 26
Population: as for outcome 1
Measure: Number; unit: unplanned visits
Arm/Group | FOM 12 mcg + FP | Fluticasone Propionate (FP)
Number analyzed (Participants) | 411 | 409
unplanned visits
  Telephone contact with study MD: V3 | 19 | 18
  Telephone contact with other MD or HCP: V3 | 5 | 9
  unplanned visit to study MD;include home:V3 | 7 | 13
  unplanned visit to other MD or HCP incl.home:V3 | 5 | 9
  Emergency or hospital visit (< 24 hours):V3 | 3 | 4
  Hospital admission or Emergency visit (>24hrs):V3 | 1 | 1
  Telephone contact with study MD: V4 | 25 | 17
  Telephone contact with other MD or HCP: V4 | 5 | 7
  unplanned visit to study MD;include home:V4 | 10 | 15
  unplanned visit to other MD or HCP incl.home:V4 | 15 | 16
  Emergency or hospital visit (< 24 hours):V4 | 3 | 4
  Hospital admission or Emergency visit (>24hrs):V4 | 0 | 2
  Telephone contact with study MD: V5 | 14 | 9
  Telephone contact with other MD or HCP: V5 | 8 | 2
  unplanned visit to study MD;include home:V5 | 6 | 9
  unplanned visit to other MD or HCP incl.home:V5 | 10 | 7
  Emergency or hospital visit (< 24 hours):V5 | 4 | 6
  Hospital admission or Emergency visit (>24hrs):V5 | 2 | 0

ADVERSE EVENTS:
Arm/Group | FOM 12 mcg + FP | Fluticasone Propionate (FP)
Serious Adverse Events (participants affected / at risk) | 10/411 | 9/409
Other Adverse Events (participants affected / at risk) | 5/411 | 9/409
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FOM 12 mcg + FP (N=411) | Fluticasone Propionate (FP) (N=409)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Dyskinesia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FOM 12 mcg + FP (N=411) | Fluticasone Propionate (FP) (N=409)
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.